CLINICAL TRIAL: NCT05059587
Title: A Randomized, Double-blind, Active-controlled, Multi-center, Phase III Study to Evaluate the Efficacy and Safety of MBA-P01 in Subjects With Moderate to Severe Glabellar Lines
Brief Title: Study to Evaluate the Efficacy and Safety of MBA-P01 in Subjects With Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medytox Korea (Industry)
Responsible Party: Sponsor
Organization: Medy-Tox (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MT14-KR20GBL309
Record Dates: First submitted 2021-09-17; First posted 2021-09-28 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2021-09

CONDITIONS: Glabellar Frown Lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MBA-P01 (Experimental): MBA-P01 will be injected into the GL: initial double-blind treatment on Day 1.
  Interventions: Drug: MBA-P01
- BOTOX® (Active Comparator): BOTOX® will be injected into the GL: initial double-blind treatment on Day 1.
  Interventions: Drug: BOTOX

INTERVENTIONS:
Drug: MBA-P01 — MBA-P01 will be injected into the Glabellar line.
  Arms: MBA-P01
Drug: BOTOX — Botox will be injected into the Glabellar line.
  Other Names: OnabotulinumtoxinA
  Arms: BOTOX®

SUMMARY:
This study is intended to evaluate the efficacy and safety of MBA-P01 compared to BOTOX in treatment of glabellar lines.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 19 and 65
* Patients attaining ≥grade 2 (moderate) in the investigator's rating of the severity of glabella lines at maximum frown
* Patients who can comply with the study procedures and visit schedule
* Patients who voluntarily sign the informed consent

Exclusion Criteria:

* Patients with medical conditions who may be at greater risk due to the administration of the investigational drugs (e.g.. diseases that may affect the neuromuscular action including Myasthenia Gravis, Lambert-Eaton Syndrome, Amyotrophic Lateral Sclerosis and motor neuropathy)
* Patients with the history of facial nerve paralysis or the symptoms of eyelid ptosis
* Patients who have received other procedures which may affect glabellar lines within 6 months
* Patients who were injected with botulinum toxin within the past 6 months
* Patients with allergy or hypersensitivity to the investigational drugs or their components
* Patients who have bleeding tendency or taking anti-coagulant
* Female subjects who are pregnant or lactating. Female subjects of childbearing age who have a plan to get pregnant during the study period, or do not use available contraceptive methods (Women of childbearing age should have negative urine pregnancy test results at baseline visit (0 week) prior to the first injection.)
* Patients with skin disorders or infection at the injection site
* Patients who are participating in other clinical trials or have participated in other clinical trials 30 days before screening
* Patients who are unable to communicate or follow the instructions
* Patients who are not eligible for this study based on the judgment of an investigator

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2021-08-30 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2022-03-29 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects achieving at least a 2-grade improvement from baseline on the facial wrinkle scale of GL at maximum frown at Week 4. | Week 4
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.

SECONDARY OUTCOMES:
Investigator-rated improvement rate of glabellar lines at maximum frown | Week 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated improvement rate of glabellar lines at maximum frown | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Investigator-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Independent photo evaluator-rated improvement rate of glabellar lines at frown | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Independent photo evaluator-rated improvement rate of glabellar lines at rest | Week 4, 8, 12, 16
  The investigator and participant evaluate the participant's GL severity using a 4-grade scale (0 to 3) where 0=none and 3 = severe.
Participant-rated satisfaction after treatment | Week 4, 8, 12, 16
  Participant evaluate the level of satisfaction by 7-grade score (1 to 7) where 1= very dissatisfied 7=very satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang Univ. Hospital, Seoul, Dongjak-gu, South Korea